CLINICAL TRIAL: NCT03698916
Title: A Multicenter Observational Study on the Use of Delivra-Celecoxib 8% Cream on Pain Experienced by Patients With Osteoarthritis of the Knees.
Brief Title: Delivra-Celecoxib 8% Cream and Osteoarthritis
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit
Sponsor: Credit Valley Rheumatology (Other)
Collaborators: Delivra, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CEL-OA-0001
Record Dates: First submitted 2018-10-02; First posted 2018-10-09 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Celecoxib cream 8% — transdermal delivery of 8% Celecoxib

SUMMARY:
This is an observation of the current use of a transdermal preparation of Celecoxib 8% which is being used in the treatment of patients with primary OA of the knees. Subjects will be followed for 12 weeks.

DETAILED DESCRIPTION:
This is an observation of the current use of a transdermal preparation of Celecoxib 8% which is being used in the treatment of patients with primary OA of the knees. This transdermal celecoxib preparation is currently in use in multiple rheumatology clinics in southern Ontario, Canada. Only patients that have been prescribed the celecoxib cream will be approached for screening and subsequent study participation. The study is purely observational as the protocol does not dictate treatment or dose assignment. Subjects will be followed for 12 weeks. In addition to the baseline clinic visit, they will participate in 2 telephone calls where data will be collected on outcome assessments that measure disease severity. The data collected during those visits will be compared to baseline values of the same assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Males or Females age 30 to 75.
2. Written informed consent
3. Patients with primary osteoarthritis (with radiological evidence) of the knees who have been prescribed Del-Cel.
4. On stable pain therapy with an oral or topical NSAID or acetaminophen.
5. Able to read and understand English to answer pain assessment questions independently.
6. Willing and able to fulfill the requirements of the study, including complete scheduled follow-up phone visits.

Exclusion Criteria:

1. Secondary OA of the study knee
2. History of pseudo gout or inflammatory flare-ups
3. Major surgery or previous damage to the study knee at any time, or minor knee surgery to the study knee within 1 year of visit 1.
4. Requires oral or intra-muscular corticosteroids or received an intra articular corticosteroid injection into the study knee within the past 90 days of visit 1, or into any other joint within the past 30 days of visit 1, or currently applying topical corticosteroids onto the study knee.
5. Received intra-articular viscosupplementation (eg, hylan G-F 20 [Synvisc®]) in the study knee in the past 6 months of visit 1.
6. On prior stable therapy (ie, more than 3 days per week for the previous month) with an opioid analgesic prior to the screening visit will be excluded.
7. Previously withdrawn from this study
8. History of fibromyalgia
9. Other painful or disabling conditions affecting the knee or leg, or disabling condition of the hands (used to apply the study drug)
10. Skin disorder with current involvement on the hands (used to apply the study drug) or the knee(s) (application site)
11. Referred to an orthopedic surgeon for consideration of, or been advised to have, knee replacement or knee reconstruction surgery
12. Radiologic evidence of OA of the knee advanced to the point that all cartilage has been eroded (ie, bone on bone)
13. Recently started using a cane within the past 30 days prior to visit 1.
14. History of chronic headaches, or other condition, that may require more than occasional use of rescue medication, e.g.: acetaminophen.

Subjects that do not meet all the enrollment criteria may not be enrolled. Any violations of these criteria must be reported in accordance with IRB Policies and Procedures.

Ages: 30 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Primary OA patients of the three rheumatology clinics included in this study protocol that have been prescribed the Delivra Celecoxib Cream 8% (Del-Cel) .
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Can study personnel enrol at least 70% of all eligible patients. | This data will be collected during recruitment. Recruitment will end when the enrolment target of 45 subjects has been met.
  The screening log will be reviewed to determine how many eligible participants consented to study participation. The evaluation may also include reasons for ineligibility. This objective will be met if the threshold of least 70% is met.
Can study personnel collect 100% of the data scheduled to be collected from at least 70% of the enrolled subjects. | Baseline data will be compared to data collected after 12-weeks of treatment.
  This objective will be met if 100% of study assessments (Western Ontario and McMaster University (WOMAC) Osteoarthritis index scores, Numeric Rating Score (NRS) Pain Index and Patient Global Assessment (PGA) score) is collected from ≥ 70% of the enrolled patients.
Calculate the Sample standard deviation of Western Ontario and McMaster University (WOMAC) Osteoarthritis index scores from this population. | Baseline data will be compared to data collected after 12-weeks of treatment.
  Higher WOMAC scores indicate an increase in disease severity, i.e.: increased pain and decrease functionality. The mean and standard deviation of the sample will be calculated from the observations collected for WOMAC assessment. It will be used for future sample size calculations.
Calculate Sample standard deviations of Patient Global Assessment (PGA) scores from this population. | Baseline data will be compared to data collected after 12-weeks of treatment.
  The standard deviations will be calculated from the observations collected for PGA. It will be used for future sample size calculations. Higher scores reflect greater disease severity from the patient's perspective. Scores range from 0- "No symptoms" to 10 "Worst symptoms imaginable"
Calculate Sample standard deviations of Numeric Rating Score (NRS) Pain Index from this population. | Baseline data will be compared to data collected after 12-weeks of treatment.
  The standard deviations will be calculated from the observations collected for NRS assessment. It will be used for future sample size calculations. Higher pain scores indicate grater pain experienced by the subject. Scores range from 0- "No pain" to 10 "Worst pain imaginable"

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Chow, MD, Principal Investigator — Credit Valley Rheumatology
Locations (3):
- Canada (3):
  - Dr. Angela Montgomery - Rheumatologist, Mississauga, Ontario
  - Dr. Brandusa Florica - Rheumatologist, Mississauga, Ontario
  - Credit Valley Rheumatology, Mississauga, Ontario

IPD SHARING:
Plan to Share IPD: No